CLINICAL TRIAL: NCT05885841
Title: Evaluation of XTR004 as a Novel 18F-labeled PET Myocardial Perfusion Imaging (MPI) Tracer in Diagnosis of Known or Suspected CAD Compared With Invasive Coronary Angiography, Fractional Flow Reserve, Index of Microcirculatory Resistance
Brief Title: Evaluation of XTR004 as a Novel 18F-labeled PET MPI Tracer in Diagnosis of Known or Suspected CAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sinotau Pharmaceutical Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STB-XTR004-201
Record Dates: First submitted 2022-12-25; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Coronary Artery Disease (CAD)
Keywords: coronary artery disease(CAD); positron emission tomography (PET)
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- XTR004 (Experimental): In the resting stage, subjects will receive an IV bolus injection of XTR004 to assess myocardial perfusion and myocardial blood flow.
  Under the pharmacological stress stage with adenosine, subjects will receive another IV bolus injection of XTR004 to assess myocardial perfusion and myocardial blood flow.
  Interventions: Drug: XTR004

INTERVENTIONS:
Drug: XTR004 — At rest: IV bolus injection of XTR004 with a dose range of 2.0-2.5 mCi
  At stress: IV infusion of adenosine at a rate of 140 μg/kg/min. IV bolus injection of XTR004 with a dose range of 6.0-7.5 mCi.

SUMMARY:
The diagnostic efficacy and safety of the XTR004 myocardial perfusion PET imaging tracer are evaluated for known or suspected CAD with the use of invasive coronary angiography as the reference standard for the diagnosis of CAD and invasive pressure-temperature FFR/IMR as a reference for the detection of abnormal coronary function.

DETAILED DESCRIPTION:
A phase II study that is single-arm, open-label, multi-center, and self-controlled with the following objectives;

1. Quantitative diagnostic efficacy of XTR004 perfusion imaging tracer in the diagnosis of known or suspected CAD using invasive coronary angiography as a reference standard for CAD.
2. The effectiveness of XTR004 myocardial perfusion imaging tracer in the detection of CAD using a pressure-temperature guide wire fractional flow reserve (FFR), and index of microcirculation resistance (IMR) as a reference standard to confirm abnormal coronary blood flow reserve and microvascular disfunction.
3. Subjects' safety after two doses of XTR004 intravenous injection.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female aged between 18 and 75 years old.
2. Symptoms associated with known or suspected CAD.
3. Having at least one risk factor for CAD, including hypertension, hyperlipidemia, diabetes, obesity, alcoholism, smoking, family history of CAD, postmenopausal women, or old age.
4. Subjects who need invasive coronary angiography and function tests based on their routine clinical examination.
5. Subjects who can understand, sign, and date the written informed consent.

Exclusion Criteria:

1. Severe cardiovascular disease, including but not limited to an acute coronary syndrome, second or third-degree atrioventricular, sinoatrial block, NYHA class iii and iv, heart failure, dilated or hypertrophic cardiomyopathy, etc., and have been assessed by the investigator as unsuitable to participate in this study.
2. Severe acute or chronic lung disease, including but not limited to chronic obstructive pulmonary disease, asthma, bronchiectasis, emphysema, pulmonary fibrosis, pulmonary embolism, pneumonia, etc., and have been assessed by the investigator as unsuitable to participate in this study.
3. Severe or unstable central nervous system disease, including but not limited to unstable cerebrovascular disease, active epilepsy, infectious disease of the central nervous system, etc., and have been assessed by the investigator as unsuitable to participate in this study.
4. Severe bleeding disorders or coagulation disorders, including but not limited to purpura, hemophilia, vitamin K deficiency, etc., and have been assessed by the investigator as unsuitable to participate in this study.
5. Severe liver disease, including but not limited to viral hepatitis, autoimmune hepatitis, liver cirrhosis, liver cancer, etc., and have been assessed by the investigator as unsuitable to participate in this study.
6. Severe renal impairment, including but not limited to glomerular nephropathy, hydronephrosis, renal cysts, etc., and have been assessed by the investigator as unsuitable to participate in this study.
7. Patients with febrile or active infectious disease, and have been assessed by the investigator as unsuitable to participate in this study.
8. Patients with serious disease of other organ systems other than those not mentioned above and have been assessed by the investigator as unsuitable to participate in this study.
9. Known to be allergic to adenosine.
10. Severe allergic reaction to alcohol.
11. Known to be allergic to iodine contrast tracers.
12. Significant occupational exposure to or treatment with ionizing radiation (e.g., more than 50 mSv/yr) within 10 years.
13. Pregnancy or lactating woman.
14. Patients with mental disorders or poor compliance.
15. Those who have participated in another clinical study 30 days before enrollment or during follow-up.
16. Men and women of reproductive age refused to adopt contraceptive plans during the study period and 6 months after the study ended.
17. Other circumstances that the investigator considers inappropriate for participating in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
Qualitative reading and semi-qualitative MPI analysis (SSS and SDS) | Day 1
  Sensitivity and specificity of XTR004 PET MPI for the detection of ≥50% and ≥70% threshold coronary stenosis.
  Sensitivity and specificity of XTR004 PET MPI for the detection of abnormal function of epicardial coronary (FFR<0.8, IMR<25), abnormal coronary microcirculation (FFR≥0.8, IMR≥25), abnormal of both (FFR<0.8, IMR≥25), and their corresponding thresholds.
Quantitative index of XTR004 PET myocardial blood flow (Stress MBF, MFR) | Day 1
  Sensitivity and specificity of XTR004 PET myocardial blood flow quantitative index (stress MBF, MFR) for the detection of ≥50% and ≥70% threshold coronary stenosis.
  Sensitivity and specificity of XTR004 PET MPI for the detection of abnormal function of epicardial coronary (FFR<0.8, IMR<25), abnormal coronary microcirculation (FFR≥0.8, IMR≥25), abnormal of both (FFR<0.8, IMR≥25), and their corresponding thresholds.

SECONDARY OUTCOMES:
Number of study participants with treatment-related adverse events as determined by safety parameter changes according to CTCAE v5.0 | 7 days post-injection
  Safety parameters included adverse events, vital signs (body temperature, blood pressure, respiration rate, pulse rate), physical examinations, laboratory tests (serum cardiac biomarkers, cardiac troponin I, serum biochemistry, haematology, and urinalysis) and electrocardiograms.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Hospital, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Beijing, Beijing Municipality